CLINICAL TRIAL: NCT05523570
Title: Phase 1, Non-randomized, Single Ascending Doses (SAD) Study Following Single Injection in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HNC364 Injectable Suspension
Brief Title: A Study to Evaluate the Safety, Tolerability, PK and PD of HNC364 Injectable Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Henovcom Bioscience Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HNC364-A101
Record Dates: First submitted 2022-08-24; First posted 2022-08-31 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 20 mg HNC364 (Experimental): pre-study will recruit 2 subjects (both male and female) to receive 20 mg HNC364 intramuscular administration to evaluate the safety and tolerability of HNC364 injectable suspension.
  Then 8 subjects will be admitted to the clinical study center on Day -1 and receive a single intramuscular dose of 20 mg HNC364 on Day 1, and undergo timed safety, PK, and PD assessments for 80 days post dose.
  Interventions: Drug: HNC364
- 40 mg HNC364 (Experimental): 8 subjects will be admitted to the clinical study center on Day -1 and receive a single intramuscular dose of 40 mg HNC364 on Day 1, and undergo timed safety, PK, and PD assessments for 29 days post dose.
  Interventions: Drug: HNC364
- 60 mg HNC364 (Experimental): 8 subjects will be admitted to the clinical study center on Day -1 and receive a single intramuscular dose of 60 mg HNC364 on Day 1, and undergo timed safety, PK, and PD assessments for 60 days post dose.
  Interventions: Drug: HNC364
- 80 mg HNC364 (Experimental): 8 subjects will be admitted to the clinical study center on Day -1 and receive a single intramuscular dose of 80 mg HNC364 on Day 1, and undergo timed safety, PK, and PD assessments for 60days post dose.
  Interventions: Drug: HNC364

INTERVENTIONS:
Drug: HNC364 — 2 subjects (both male and female) to receive 20 mg HNC364 intramuscular administration to evaluate the safety and tolerability of HNC364 injectable suspension. Then 8 subjects are planned for enrollment in each cohort (the ratio of male to female is as close as possible) to receive 20 mg HNC364 intramuscular administration. The proposed dose levels for use were determined to be appropriate based on the collective nonclinical data (pharmacology and toxicology) for HNC364 and the nonclinical and clinical data of the marketed drug rasagiline.
  Other Names: HNC364 injectable suspension
  Arms: 20 mg HNC364
Drug: HNC364 — 8 subjects are planned for enrollment in each cohort (the ratio of male to female is as close as possible) to receive 40 mg HNC364 intramuscular administration. The proposed dose levels for use were determined to be appropriate based on the collective nonclinical data (pharmacology and toxicology) for HNC364 and the nonclinical and clinical data of the marketed drug rasagiline.
  Other Names: HNC364 injectable suspension
  Arms: 40 mg HNC364
Drug: HNC364 — 8 subjects are planned for enrollment in each cohort (the ratio of male to female is as close as possible) to receive 60 mg HNC364 intramuscular administration. The proposed dose levels for use were determined to be appropriate based on the collective nonclinical data (pharmacology and toxicology) for HNC364 and the nonclinical and clinical data of the marketed drug rasagiline.
  Other Names: HNC364 injectable suspension
  Arms: 60 mg HNC364
Drug: HNC364 — 8 subjects are planned for enrollment in each cohort (the ratio of male to female is as close as possible) to receive 80 mg HNC364 intramuscular administration. The proposed dose levels for use were determined to be appropriate based on the collective nonclinical data (pharmacology and toxicology) for HNC364 and the nonclinical and clinical data of the marketed drug rasagiline.
  Other Names: HNC364 injectable suspension
  Arms: 80 mg HNC364

SUMMARY:
This is a non-randomized, dose-escalation first-in-human study to evaluate the safety, tolerability, PK, and PD of HNC364 following intramuscular administration of single ascending doses.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet any of the following criteria must be excluded from the study:

1. Prior to screening, subjects had clinically significant disease history as determined by the Investigator, including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immunological, psychiatric, cardio cerebrovascular disease or any reported history of sleep disorder.2. Any history of suicide or at high risk for suicide assessment at screening.

3. The subject has a history of severe allergy or allergy to the the study drug and any of its components or related excipients.

4. Prior to screening, those who have a history of gastrointestinal, liver and kidney diseases or surgery that potentially affect the absorption, distribution, metabolism and excretion of the study drug (except for uncomplicated appendectomy and hernia repair).

5. A history of alcoholism (alcoholism is defined as drinking 14 units of alcohol per week: 1 unit = 285 ml of beer, 25 ml of spirits, or 100 ml of wine) or positive alcohol breath test during the screening period.

6. Those who had a history of drug abuse or used drugs within 2 years before screening or those who were positive for urinary drug screening during the screening period.

7. Subjects who had a history of smoking or used other nicotine-containing products within 3 months before the study drug administration, or who were positive for urine nicotine test during screening.

8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.

9. Strong inhibitors and/or inducers of liver metabolizing enzymes (CYP1A2, 2A6, 2C8, 2C19, 3A4 and 3A5), strong inhibitors of liver metabolizing enzymes such as ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, acerbicin, etc., and strong inducers of liver metabolizing enzymes such as rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc. were used within 4 weeks before the study drug administration.

10. Any prescription drug, over-the-counter drug, any vitamin product or Chinese herbal medicine used within 2 weeks before the study drug administration.

11. Had consumed a special diet (including pitaya, mango, grapefruit, or certain foods containing high amounts of tyramine, etc.) or had vigorous exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc., within 2 weeks before the administration.

12. Had consumed chocolate, any food or beverage containing caffeine or xanthine-rich within 72 hours before the study drug administration.

13. Taking any alcoholic product within 48 hours before the administration. 14. Donation of plasma within 30 days, or donation of blood or massive blood loss (≥ 400 ml) within 60 days, or donation of bone marrow or peripheral stem cells within 90 days before the study drug administration.

15. Participated in other clinical trials within 30 days prior to study drug administration.

16. Acute disease or concomitant medication from the signing of informed consent form to the study drug administration.

17. Lactating women or those with positive serum pregnancy results. 18. The researchers believe that subjects with other factors that are not suitable to participate in this study.

Prohibitions and Restrictions：

1. Subjects must be willing to adhere to the following prohibitions and restrictions during the study (until final discharge from the clinic):
2. Use of tobacco- or nicotine-containing products, in any form, is prohibited within 3 months prior to study drug administration on Day 1 until after the EOS visit.
3. Within 4 weeks prior to study drug administration until 30 days post dose, any drugs known to strongly inhibit and/or induce metabolizing enzymes (CYP1A2, 2A6, 2c8, 2c19, 3A4 and 3A5) are contraindicated for use with HNC364, strong inhibitors of liver metabolizing enzymes
4. Within 4 weeks prior to study drug administration until 30 days post dose, dextromethorphan is contraindicated for use with HNC364.
5. Within 2 weeks prior to study drug administration until 44 days post dose, Meperidine, tramadol, methadone, propoxyphene, and MAO inhibitors (MAOIs), including other selective MAO-B inhibitors are contraindicated for use with HNC364.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events | Day 1 to 80 days post dose
  This safety outcome lists the number of subjects experiencing adverse events (AEs), whether not related, possibly or unlikely related to the study treatment.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Time to maximum concentration (Tmax) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Time at which half the drug has been eliminated (t½) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Area under the concentration-time curve (AUC) from time 0 to the last measurable concentration (AUC0-last) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
AUC extrapolated to infinity (AUC0-inf) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Mean residence time (MRT) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Apparent total clearance for extravascular administration (CL/F) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Apparent volume of distribution during terminal phase (Vz/F) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Elimination rate constant (Kel) | Day 1 to 80 days post dose
  PK blood samples will be collected at the following timepoints: pre dose (within 60 min); post dose at 1, 4, 8, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.
Platelet MAO-B activity | Day 1 to 80 days post dose
  Blood samples for PD analysis will be collected at the same following timepoints: pre dose (within 60 min); post dose at 4, 12 (±5 min), 24, 48, 72, 96, 120 and 144 h (±60 min); Days 9, 11, 13, 15, 17, 20, 23, 26, 29, 34, 39, 46, 53, 60, 70 and 80.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, MD, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No